CLINICAL TRIAL: NCT01129856
Title: Evaluation of Dexamethasone Phosphate Delivered by Ocular Iontophoresis for the Treatment of Dry Eye in the Controlled Adverse Environment (CAE) Model
Brief Title: Safety and Efficacy Study of EGP-437 (Dexamethasone Phosphate Formulated for Ocular Iontophoresis) to Treat Dry Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eyegate Pharmaceuticals, Inc. (Industry)
Responsible Party: Stephen From / President and Chief Executive Officer, Eyegate Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EGP-437-003
Record Dates: First submitted 2010-05-20; First posted 2010-05-25 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-04

CONDITIONS: Dry Eye
Keywords: Dry eye; Keratoconjunctivitis sicca; Iontophoresis; Ophthalmic drug delivery; EGP-437; Dexamethasone phosphate
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ocular Iontophoresis EGP-437, Low Dose (Active Comparator): Ocular Iontophoresis with EGP-437 4.0 mA-min at 1.5 mA
  Interventions: Drug: Dexamethasone phosphate ophthalmic solution
- Ocular Iontophoresis EGP-437, High Dose (Active Comparator): Ocular Iontophoresis with EGP-437 6.5 mA-min at 2.5 mA
  Interventions: Drug: Dexamethasone phosphate ophthalmic solution
- Ocular Iontophoresis Placebo (Placebo Comparator): Ocular Iontophoresis with Placebo 6.5 mA-min at 2.5 mA
  Interventions: Drug: Sodium citrate buffer solution

INTERVENTIONS:
Drug: Dexamethasone phosphate ophthalmic solution — Transscleral iontophoresis delivery of EGP-437 (dexamethasone phosphate formulated for ocular iontophoresis)
  Arms: Ocular Iontophoresis EGP-437, High Dose; Ocular Iontophoresis EGP-437, Low Dose
Drug: Sodium citrate buffer solution — Sodium citrate buffer solution 100 mM
  Arms: Ocular Iontophoresis Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of EGP-437 (dexamethasone phosphate formulated for ocular iontophoresis) using the EyeGate® II Iontophoresis system in patients with dry eye.

DETAILED DESCRIPTION:
Dry eye is the most prevalent form of ocular discomfort and irritation. Estimates range from 20 million people in the United States being affected with mild to moderate dry eye, to as many as one out of every five Americans.

EyeGate completed a single-center, randomized, double-masked, placebo-controlled Phase 2 efficacy study in 105 subjects with mild to moderate dry eye disease, utilizing the Controlled Adverse Environment (CAE), a clinical model which allows for standardized measurement of dry eye signs and symptoms in the investigation of therapeutic agents. In this Phase 2 study, the improvements documented in dry eye signs and symptoms relative to the placebo group indicated that the ocular iontophoresis treatments with EGP-437 (dexamethasone phosphate formulated for ocular iontophoresis) had both a rapid onset of action and a long-term effectiveness.

The Phase 3 study is intended to confirm and extend the results from the Phase 2 study, utilizing the CAE model. The study is designed to assess the safety and efficacy of EGP-437 at two different dose levels: Ocular Iontophoresis with EGP-437 4.0 mA-min at 1.5 mA and Ocular Iontophoresis with EGP-437 6.5 mA-min at 2.5 mA compared to Ocular Iontophoresis with placebo (sodium citrate buffer solution) for the treatment of the signs and symptoms of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Have a reported history of dry eye in each eye
* Be at least 12 years of age
* Demonstrate a response when exposed to the Controlled Adverse Environment model at Visits 1 and 2

Exclusion Criteria:

* Have contraindications to the use of the test articles
* Have known allergy or sensitivity to the study medications or their components
* Have any ocular infections, active ocular inflammation, or preauricular lymphadenopathy
* Be current contact lens wearers or wear contacts during the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2010-06; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Sign: Differences in corneal fluorescein staining (inferior region, Ora Scale) Visit 1 Pre-CAE to Visit 6 compared to placebo; Symptom: Ocular discomfort at Visit 5 as compared to placebo | Up to 10 weeks

SECONDARY OUTCOMES:
Sign: Corneal fluorescein staining (each region, Ora Scale); Symptom: Ocular discomfort pre- and post-CAE (Ora Scale) | Up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gail L Torkildsen, MD, Principal Investigator — Andover Eye Associates
Locations (5):
- United States (5):
  - The Eye Care Group, Waterbury, Connecticut
  - Central Maine Eye Care, Lewiston, Maine
  - Andover Eye Associates, Andover, Massachusetts
  - Total Eye Care, Memphis, Tennessee
  - Virginia Eye Consultants, Norfolk, Virginia